CLINICAL TRIAL: NCT05351385
Title: S Protein and COVID-19: a Monocentric Prospective Study
Acronym: PROS-Covid
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Milano Bicocca (Other)
Collaborators: San Gerardo Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PROS-Covid
Record Dates: First submitted 2021-10-05; First posted 2022-04-28 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: COVID-19
Keywords: PROS; S Protein; SARS-CoV-2; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Real-Time Polymerase Chain Reaction; Bronchoalveolar Lavage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Nasopharyngeal swab, Bronchoalveolar lavage, Peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Covid +: Patients SARS-CoV-2 positive.
  Interventions: Procedure: Hematolgy and Chemistry analysis; Procedure: Real Time PCR; Procedure: PROS assay COVID+; Procedure: Sflt1 assay COVID+
- Control: Patients with Pneumonia non-SARS-CoV-2 related
  Interventions: Procedure: PROS assay CONTROL; Procedure: Sflt1 assay CONTROL

INTERVENTIONS:
Procedure: Hematolgy and Chemistry analysis — Samples will be collected at Day 0, Day 5, Day 10 and Day 15
  Other Names: Peripheral Blood
  Groups: Covid +
Procedure: Real Time PCR — Samples will be collected at Day 0, Day 5, Day 10 and Day 15
  Other Names: Nasopharyngeal swab; Bronchoalveolar lavage
  Groups: Covid +
Procedure: PROS assay COVID+ — Samples will be collected at Day 0, Day 5, Day 10 and Day 15
  Other Names: Peripheral Blood
  Groups: Covid +
Procedure: Sflt1 assay COVID+ — Samples will be collected at Day 0 and Day 10
  Other Names: Peripheral Blood
  Groups: Covid +
Procedure: PROS assay CONTROL — Samples will be collected at Day 0 (+5)
  Other Names: Peripheral Blood
  Groups: Control
Procedure: Sflt1 assay CONTROL — Samples will be collected at Day 0 (+5)
  Other Names: Peripheral Blood
  Groups: Control

SUMMARY:
The aim of this study is to compare plasma S Protein levels to SARS-CoV-2 viral load in COVID positive patients.

DETAILED DESCRIPTION:
Non-pharmacological, non-interventional, prospective, monocentric study involving the use of biological materials.

There will be two cohorts:

* COVID + cohort: 50 patients with positive nasopharyngeal swab and / or BAL.
* Control Cohort: 20 patients with non-SARS-CoV-2 related pneumonia.

The study involves analyzing biological samples collected for normal clinical practice.

In particular:

* blood samples will be used for PROS and Sflt1 assay, haematological, biochemical and coagulation tests.
* Samples deriving from nasopharyngeal swab or from Broncho-Alveolar Lavage (BAL) liquid will be used for Real time PCR analysis to evaluate the viral load of SARS CoV-2.

ELIGIBILITY:
Inclusion Criteria:

Cohort COVID + :

* Subjects aged ≥ 18 years.
* Signing of the informed consent.
* Positivity for SARS-CoV-2 by RealTimePCR from nasopharyngeal swab or bronchial wash.

Cohort Control:

1. Subjects aged ≥ 18 years.
2. Signing of the informed consent.
3. Diagnosis of pneumonia not related to SARS-CoV-2, demonstrated by negative swab.

Exclusion Criteria:

* Patients with a diagnosis of congenital S Protein deficiency.
* Patients who are taking oral anticoagulant therapy (TAO) or new oral anticoagulants (NAO).
* Chronic liver failure (> 5 points on the Child-Pugh score).
* Female subjects who are pregnant or on estrogen-progestogen replacement therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Pneumonia SARS-CoV-2 related or not related
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-09-23 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2024-12-03 (Estimated)

PRIMARY OUTCOMES:
Plasma PROS levels compared to early stage of SARS-CoV-2 infection. | Day 0
  To demonstrate a correlation between low plasma PROS levels and the early stage of SARS-CoV-2 infection, defined as the first 10 days after onset of symptoms.
Plasma PROS levels compared to early stage of SARS-CoV-2 infection. | Day +5
  To demonstrate a correlation between low plasma PROS levels and the early stage of SARS-CoV-2 infection, defined as the first 10 days after onset of symptoms.
Plasma PROS levels compared to early stage of SARS-CoV-2 infection. | Day +10
  To demonstrate a correlation between low plasma PROS levels and the early stage of SARS-CoV-2 infection, defined as the first 10 days after onset of symptoms.
Plasma PROS levels compared to early stage of SARS-CoV-2 infection. | Day +15
  To demonstrate a correlation between low plasma PROS levels and the early stage of SARS-CoV-2 infection, defined as the first 10 days after onset of symptoms.
Plasma PROS level compared to SARS-Cov-2 viral load | Day 0
  To demonstrate a correlation between PROS and the viral load of SARS-CoV-2
Plasma PROS level compared to SARS-Cov-2 viral load | Day+5
  To demonstrate a correlation between PROS and the viral load of SARS-CoV-2
Plasma PROS level compared to SARS-Cov-2 viral load | Day+10
  To demonstrate a correlation between PROS and the viral load of SARS-CoV-2
Plasma PROS level compared to SARS-Cov-2 viral load | Day+15
  To demonstrate a correlation between PROS and the viral load of SARS-CoV-2

SECONDARY OUTCOMES:
Normal plasma protein S levels in patients with Pneumonia non-SARS-CoV related | Day 0, Day +5
  To confirm the non-consumption of protein S in Pneumonia other than SARS-CoV-2.
Normal levels Plasma S potein in late stage of SARS-CoV-2 infection in COVID + patients. | Day 0, Day +5, Day +10, Day+15
  To confirm normalization of plasma S Potein levels longitudinally during the late stages of SARS-CoV-2 infection.
Correlation between plasma levels of S protein and the severity indices of SARS-CoV-2 disease | Day 0, Day +5, Day +10, Day+15
  To detect any correlations between plasma levels of S Protein and already known parameters indicative of SARS-CoV-2 disease severity (e.g. days spent in O2 at high flows or the need for intubation; access to the Intensive Care Unit; appearance of arterial or venous thromboembolic events; coagulation activation markers; markers of inflammatory or cytokine phase; mortality).
Plasma protein S as an index for use of immunosuppressive therapy. | Day 0, Day +5, Day +10, Day+15
  To use protein S values as an indicator for the introduction of immunosuppressive drugs in therapy in patients with COVID-19 disease.

CONTACTS AND LOCATIONS:
Overall Officials: Luisa Verga, MD, Study Director — San Gerardo Hospital
Locations (1):
- San Gerardo Hospital, Monza, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No